CLINICAL TRIAL: NCT05894655
Title: CO-CREATE-Ex: Community-engaged Optimization of COVID-19 Rapid Evaluation And TEsting Experiences
Brief Title: Community-engaged Optimization of COVID-19 Rapid Evaluation And TEsting Experiences
Acronym: CO-CREATE-Ex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: San Ysidro Health Center (Other)
Responsible Party: Principal Investigator, Louise Laurent, MD/PhD, Principal Investigator, University of California, San Diego
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 806121
Record Dates: First submitted 2023-03-02; First posted 2023-06-08 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: COVID-19; COVID-19 Pandemic
Keywords: covid-19 testing; vaccine hesitancy; implementation; vending machine
MeSH Terms: conditions — COVID-19; Vaccination Hesitancy | interventions — Community Health Workers

STUDY DESIGN:
Intervention Model Description: The investigators chose a roll-out implementation optimization (ROIO) design to implement the study. This is a novel implementation science study design that affords a balance of rigor and flexibility to rapidly and iteratively refine in response to dynamic contexts like the pandemic.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- San Ysidro Health Center - Main Clinic (Placebo Comparator): At the main clinic all 3 strategies will be available: walk-up testing, vending machine, and Community Health Worker (CHW) providing education.
  Interventions: Behavioral: COVID-19 walk-up, on-site testing strategy; Behavioral: Community Health Worker (CHW) leading testing navigation and general preventive care reminders; Behavioral: No-cost self-testing kit vending machines
- San Ysidro Health Center - Logan Heights (Experimental): A vending machine and Community Health Worker (CHW) providing education will be available at Logan Heights
  Interventions: Behavioral: Community Health Worker (CHW) leading testing navigation and general preventive care reminders; Behavioral: No-cost self-testing kit vending machines
- San Ysidro Health Center - Lincoln Park (Experimental): A vending machine and Community Health Worker (CHW) providing education will be available at Lincoln Park
  Interventions: Behavioral: Community Health Worker (CHW) leading testing navigation and general preventive care reminders; Behavioral: No-cost self-testing kit vending machines
- San Ysidro Health Center - Chula Vista (Experimental): A vending machine and Community Health Worker (CHW) providing education will be available at Chula Vista
  Interventions: Behavioral: Community Health Worker (CHW) leading testing navigation and general preventive care reminders; Behavioral: No-cost self-testing kit vending machines

INTERVENTIONS:
Behavioral: COVID-19 walk-up, on-site testing strategy — This strategy is a no-appointment, walk-up point-of-care PCR and rapid testing strategy for clinic patients and community members. It will be offered 5 days/week for 7 hours during the first 3 months of the trial at Clinic 1. The intensity will decrease over the trial ending with 1 SYH Medical Assistant overseeing the testing protocol. Bilingual research staff will be trained to oversee onsite testing.
  Arms: San Ysidro Health Center - Main Clinic
Behavioral: Community Health Worker (CHW) leading testing navigation and general preventive care reminders — This strategy provides health counseling about when COVID-19 testing is recommended, which test to use, testing instructions, and how to interpret results. Community Health Workers (CHW) will also offer general preventive health care reminders such as flu shots, blood pressure checks, and A1c screenings. This strategy will be available full-time during the first 3 months of roll-out at each clinic and after 3 months, the CHW will be available as needed. Trained bilingual CHW will be supervised by a SYH employee.
Behavioral: No-cost self-testing kit vending machines — This strategy includes vending machines that will provide interactive instructions for accessing free self-testing COVID-19 kits located outside of clinics for patients and community members to use anytime. The vending machines will be available 24 hours/day, 7 days a week.

SUMMARY:
Throughout the Coronavirus disease (COVID-19) pandemic, rates of COVID-19 have been persistently high in San Diego County's central and southern communities near the United States/Mexico border. These regions predominantly house Latino residents, the ethnic minority community most impacted by COVID-19 in San Diego. In the Phase I project, University of California, San Diego (UCSD) partnered with San Ysidro Health (SYH) and the Global Action Research Center, to co-create and demonstrate the impact of a COVID-19 testing program in San Ysidro, one of the most impacted areas from COVID-19 in San Diego County. To date, the project tested >10,000 community members (92% Latino) and received requests to scale-out the testing program to additional primary care clinic sites.

In this Phase III project, Community-engaged Optimization of COVID-19 Rapid Evaluation And TEsting Experiences (CO-CREATE-Ex) will extend work with the Phase I community and clinical partners to refine, specify, implement, and evaluate an implementation strategy bundle that optimizes COVID-19 testing, expanding beyond current polymerase chain reaction (PCR) testing to FDA-authorized COVID-19 rapid antigen testing.

DETAILED DESCRIPTION:
CO-CREATE-Ex will roll-out our implementation using 3 strategies:

1. keeping the current, walk-up free testing protocol
2. Offering Community Health Worker (CHW) to lead COVID-19 test counseling, preventive care reminders, and offer testing support
3. Installing vending machines that will dispense FDA-authorized self-testing kits.

For each strategy, participants will consent into study, provide demographics and test history, and receive a free rapid antigen test (RAT) kit. After receiving the test kit, participants will be prompted to return their results and fill out a survey about their COVID-19 experiences. Study subjects will be contacted up to three times over a course of 4 weeks to return their results and complete the survey. Study coordinators will use participants' preferred method of contact.

ELIGIBILITY:
Inclusion Criteria:

* Speak English and/or Spanish
* Affiliated with San Ysidro Health as a patient at select clinics (San Ysidro, Chula Vista, Lincoln Park, and Logan Heights) OR
* A member of a community near a San Ysidro Health clinic (San Ysidro, Chula Vista, Lincoln Park, and Logan Heights).

Exclusion Criteria:

* Institutionalization for psychiatric disorder, developmental delay, or criminal activity.
* Unable to provide informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6527 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
Identify solutions and evaluation methods to refine a multi-component implementation strategy bundle using a Community and Scientific Advisory Board. | 2 years
  The primary objective is to refine and operationalize the multi-component implementation strategy bundle and measures of implementation and sustainment success for rapid FDA-authorized COVID-19 rapid testing using the partnership with the Global Arc and Community and Scientific Advisory Board. Each session will be recorded while Global Arc partners guide the board to identify potential failures in the implementation design. Measures of success will be collected by partner engagement surveys, which will be administered and analyzed after each meeting.

SECONDARY OUTCOMES:
Number of distributed rapid antigen tests within our target communities as measured by a proxy outcome. | 18 months
  The secondary objective is to implement and evaluate the impact of our multicomponent implementation strategy bundle to optimize COVID-19 rapid testing among underserved, Latino communities. Implementation strategies include a vending machine, Community Health Workers, and walk-up testing tables. Each strategy will be rolled-out across four clinics over 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Laurent, MD/PhD, Principal Investigator — University of California, San Diego
Locations (1):
- San Ysidro Health Centers, San Ysidro, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salgin L, Reyes BJ, Bojorquez MB, Lomeli A, Velasquez S, Cain KL, Seifert M, Laurent LC, Stadnick NA, Rabin BA. Using multi-method approaches to document and assess adaptations in a community-driven COVID-19 testing program. Implement Sci Commun. 2026 Feb 5. doi: 10.1186/s43058-026-00871-9. Online ahead of print. PMID 41639712
- [Derived] Stadnick NA, Laurent LC, Cain KL, Seifert M, Burola ML, Salgin L, Watson P, Oswald W, Munoz FA, Velasquez SF, Smith JD, Zou J, Rabin BA. Community-engaged optimization of COVID-19 rapid evaluation and testing experiences: roll-out implementation optimization trial. Implement Sci. 2023 Oct 2;18(1):46. doi: 10.1186/s13012-023-01306-y. PMID 37784200